CLINICAL TRIAL: NCT04308421
Title: A Prospective, Double-blind, Split-body, Randomized Controlled Trial to Assess the Efficacy of Low Level Laser Therapy for Pigmentary Disorders
Brief Title: Efficacy of Red Light in the Treatment of Pigmentary Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Sunil Kalia, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H20-00293
Record Dates: First submitted 2020-02-25; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Melasma; Lichen Planus Pigmentosus; Vitiligo
Keywords: Melasma; Lichen planus pigmentosus; Vitiligo; Low level laser therapy; Photobiomodulation; Red light; Pigmentation disorders
MeSH Terms: conditions — Melanosis; Vitiligo; Pigmentation Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Low level red light/laser (Experimental): Patients will be treated twice a week for 12 weeks with low irradiation 650 nm +/- 5 nm red light on one randomly allocated side of the face or body
  Interventions: Device: Red light
- Control side (No Intervention): An affected area on the contralateral side of the face or body or within a single patch will not be treated

INTERVENTIONS:
Device: Red light — Low irradiation 650 nm +/- 5 nm red light
  Other Names: Low level laser therapy
  Arms: Low level red light/laser

SUMMARY:
Pigmentary disorders such as melasma, lichen planus pigmentosus and vitiligo can significantly affect patients' quality of life. Treatment responses are usually slow and typically have limited efficacy. In recent years, low level laser therapy has been an emerging treatment modality for androgenetic alopecia, acne, wound healing and photorejuvenation. This is a prospective, double-blind, split-body, randomized controlled trial assessing the efficacy of low level laser therapy with red light for pigmentary disorders such as, melasma, lichen planus pigmentosus and vitiligo.

DETAILED DESCRIPTION:
This will be a participant and evaluator blinded trial with random allocation of one side of the face or affected area to treatment and the contralateral side as control. Random allocation of the treatment side will be performed using randomization software. Participants will be treated twice a week for 12 weeks with low irradiation 650 nm +/- 5 nm red light and followed up 4 weeks after completion of treatment. A trained blinded evaluator will assess clinical outcomes on week 4, week 8, week 12 and at follow up at week 16, using validated scores.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older.
* Participants should be competent to give fully informed consent by themselves
* Should have received a diagnosis of either melasma, lichen planus pigmentosus or vitiligo either clinically or pathologically and have bilateral facial hyperpigmentation/depigmentation or bilateral similar sized depigmented/hyperpigmented patches or a single patch larger than 25 cm2.
* Participants must stop receiving topical treatments or phototherapy 4 weeks prior to commencing the study

Exclusion Criteria:

* Known photosensitivity disorder
* Unable to attend follow up appointments or twice weekly treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in Modified-MASI (Melasma Area and Severity Index) compared to baseline for melasma and lichen planus pigmentosus | Week 0, week 4, week 8, week 12 and at follow up at week 16
  A trained blinded evaluator will assess clinical outcomes on week 4, week 8, week 12 and at follow up at week 16, using validated scores to assess change from baseline
Change in DPASI (Dermal Pigmentation Area and Severity score) compared to baseline for lichen planus pigmentosus | Week 0, week 4, week 8, week 12 and at follow up at week 16
  A trained blinded evaluator will assess clinical outcomes on week 4, week 8, week 12 and at follow up at week 16, using validated scores to assess change from baseline
Change in VASI (Vitiligo Area Scoring Index) compared to baseline for vitiligo | Week 0, week 4, week 8, week 12 and at follow up at week 16
  A trained blinded evaluator will assess clinical outcomes on week 4, week 8, week 12 and at follow up at week 16, using validated scores to assess change from baseline

SECONDARY OUTCOMES:
Colorimeter measurements | Week 0, week 4, week 8, week 12 and at follow up at week 16
  Change in average L*a*b color system will be measured for background skin and the area of hyperpigmentation or depigmentation from baseline.

OTHER OUTCOMES:
Physician Global Assessment | Week 16
  Physician global assessment at the end of treatment at follow up will be assessed to identify change in pigmentation compared to baseline photographs.
Patient global assessment | Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- The Skin Care Centre, Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No